CLINICAL TRIAL: NCT04815681
Title: Evaluating an Online Single-session Intervention for Mental Health and Wellness of Greek Adolescents
Brief Title: Evaluating an Online Wellness Intervention for Greek Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll participants
Sponsor: University of Pennsylvania (Other)
Collaborators: National and Kapodistrian University of Athens, Greece (Unknown); University Mental Health, Neurosciences and Precision Medicine Research Institute "Costas Stefanis," Greece (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 844481
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Depressive Symptoms; Anxiety; Happiness
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Elements Toolbox (COMET) (Experimental)
  Interventions: Behavioral: Common Elements Toolbox
- Active Control Condition (Active Comparator)
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Common Elements Toolbox — COMET is an online unguided self-help intervention that lasts approximately 40-50 minutes.
  Other Names: COMET
  Arms: Common Elements Toolbox (COMET)
Behavioral: Active Control — The active control condition includes an online self-awareness program that lasts approximately 40-50 minutes. Participants in the control condition will receive access to the intervention after data collection for the study has been completed.
  Arms: Active Control Condition

SUMMARY:
The investigators are evaluating the effects of an online single-session mental health intervention (the Common Elements Toolbox; COMET). To evaluate COMET, the investigators are conducting a randomized controlled trial with Greek adolescents attending high school in the Attica region in Greece. Students will be randomized to the COMET condition or to an active control condition.

Primary outcome measures (depressive symptoms, anxiety symptoms, subjective well-being) will be measured at two weeks post-intervention and four weeks post-intervention.

The investigators will evaluate COMET as a universal intervention (using the full sample) and as a targeted intervention (analyzing those who reported elevated depressive symptoms or anxiety symptoms at baseline).

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 20 years old and a student at a participating Greek high school. Access to the internet.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-8 (PHQ-8) | Up to 4 weeks post-intervention
  Depression questionnaire. Scores range from 0 to 24. Lower scores indicate less depression.
Change in Generalized Anxiety Disorder Screener-7 (GAD-7) | Up to 4 weeks post-intervention
  Anxiety questionnaire. Total scores range from 0-21. Lower scores indicate less anxiety.
Change in the Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | Up to 4 weeks post-intervention
  Subjective Well-being questionnaire. Total scores range from 7 to 35. Higher values indicate higher well-being scores.

SECONDARY OUTCOMES:
Ratings on the Acceptability of Intervention Measure (AIM) | Immediately after the intervention
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate higher acceptability ratings.
Ratings on the Intervention Appropriateness Measure (IAM) | Immediately after the intervention
  Questionnaire measuring the appropriateness of an intervention. Appropriateness refers to the perceived fit or relevance of an intervention. The total score ranges from 4 to 20. Higher scores indicate higher appropriateness.
Secondary Control | Up to 4 weeks post-intervention
  The investigators will ask participants three items to assess secondary control (Weisz et al., 2010). The items are scored on a 4-point Likert scale, ranging from 0 ("Very false") to 3 ("Very true"). The three items are: When something bad happens, I can find a way to think about it that makes me feel better. After a really hard day, I can make myself feel better by remembering some good things that happened. When bad things happen to me that I can't control, there are lots of things I can do to feel better. Higher scores indicate greater secondary control.
Perceived Utility | Immediately after intervention
  Participants will be asked to rate three items relating to the perceived utility of each module. Specifically, the investigators asked participants: How helpful the module was; How engaging the module was; How much they will continue applying content from the module. If items are at least moderately correlated (r > .5) the investigators will combine them in a single measure of perceived utility. Higher scores indicate greater perceived utility.
Positive and Negative Affect Schedule (PANAS) | Up to 4 weeks post-intervention
  Questionnaire measuring positive affect and negative affect. Scores on the positive affect subscale range from 10-50, with higher scores representing higher levels of positive affect. Scores on the negative affect subscale range from 10-50, with lower scores representing lower levels of negative affect.

CONTACTS AND LOCATIONS:
Locations (2):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Eginition Hospital National and Kapodistrian University of Athens School of Medicine, Athens, Greece

IPD SHARING:
Plan to Share IPD: No